CLINICAL TRIAL: NCT02921230
Title: A Randomized Trial Comparing the ELUVIA Drug-eluting Stent Versus Bare Metal Self-expanding Nitinol Stents in the Treatment of Superficial Femoral and/or Proximal Popliteal Arteries
Brief Title: Trial Comparing ELUVIA Versus Bare Metal Stent in Treatment of Superficial Femoral and/or Proximal Popliteal Artery
Acronym: EMINENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2366
Record Dates: First submitted 2016-09-06; First posted 2016-10-03 (Estimated); Results first posted 2024-10-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Arterial Occlusive Diseases; Atherosclerosis; Vascular Diseases; Arteriosclerosis
Keywords: atherosclerosis; Superficial Femoral Artery (SFA); Proximal Popliteal Artery (PPA); stenting; paclitaxel
MeSH Terms: conditions — Arterial Occlusive Diseases; Atherosclerosis; Vascular Diseases; Arteriosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ELUVIA Stent Implantation (Experimental): Peripheral stenting
  Interventions: Device: Peripheral stenting
- control Bare Metal Stent Implantation (Active Comparator): Peripheral stenting
  Interventions: Device: Peripheral stenting

INTERVENTIONS:
Device: Peripheral stenting — stent implantation during the index procedure

SUMMARY:
The EMINENT study is a prospective, multi-center study evaluating the effectiveness of the ELUVIA stent versus Self-Expanding Bare Nitinol Stents in the treatment of lesions in the femoropopliteal arteries.

DETAILED DESCRIPTION:
The EMINENT study is a prospective, multi-center study evaluating the effectiveness of the ELUVIA stent versus Self-Expanding Bare Nitinol Stents in the treatment of lesions 30-210 mm long located in the femoropopliteal arteries in subjects with symptoms classified as Rutherford categories 2-4.

The study is a 2:1 randomized (ELUVIA vs Self-Expanding Bare Nitinol Stents), controlled, single-blind, superiority trial (RCT).

The objective of the study is to evaluate the effectiveness of the ELUVIA Drug-Eluting Vascular Stent System (ELUVIA Stent) for treating Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) lesions up to 210 mm in length when compared against bare metal stents, and collect additional data including health economics data.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 and older
2. Subject is willing and able to provide consent before any study-specific test or procedure is performed, signs the consent form, and agrees to attend all required follow-up visits
3. Chronic, symptomatic lower limb ischemia defined as Rutherford categories 2, 3 or 4
4. Stenotic, restenotic or occlusive lesion(s) located in the native Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA):

   1. Degree of stenosis ≥ 70 % by visual angiographic assessment
   2. Vessel diameter ≥ 4 and ≤ 6 mm
   3. Total lesion length (or series of lesions) ≥ 30 mm and ≤210 mm (Note: Lesion segment(s) must be fully covered with one or two overlapping ELUVIA stent(s) or Self Expanding Bare Nitinol stent(s))
   4. For occluded lesions (chronic occlusions) requiring use of re-entry device, lesion length ≤ 180 mm
   5. Target lesion located at least three centimeters above the inferior edge of the femur
5. Patent infrapopliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (< 50 % stenosis) to the ankle or foot with no planned intervention

Exclusion Criteria:

1. Previously stented target lesion/vessel
2. Target lesion/vessel previously treated with drug-coated balloon within 12 months prior to randomization/enrollment
3. Subjects who have undergone prior surgery of the SFA/PPA in the target limb to treat atherosclerotic disease
4. Use of atherectomy, laser or other debulking devices such as Rotarex in the target limb SFA/PPA during the index procedure
5. History of major amputation in the target limb
6. Documented life expectancy less than 24 months due to other medical co-morbid condition(s) that could limit the subject's ability to participate in the clinical study, limit the subject's compliance with the follow-up requirements, or impact the scientific integrity of the clinical study
7. Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated
8. Known hypersensitivity/allergy to the stent system or protocol related therapies (e.g., nitinol, paclitaxel, or structurally related compounds, polymer or individual components, and antiplatelet, anticoagulant, thrombolytic medications)
9. Platelet count less than 80000 mm3 or more than 600000 mm3 or history of bleeding diathesis
10. Concomitant renal failure with a serum creatinine higher than 2.0 mg/dL
11. Receiving dialysis or immunosuppressant therapy
12. History of myocardial infarction (MI) or stroke/cerebrovascular accident (CVA) within 6 months prior to randomization/enrollment
13. Unstable angina pectoris at the time of randomization/enrollment
14. Pregnant, breast feeding, or plan to become pregnant in the next 5 years
15. Current participation in an investigational drug or device clinical study that has not completed the primary endpoint at the time of randomization/ enrollment or that clinically interferes with the current study endpoints (Note: studies requiring extended follow-up for products that were investigational, but have become commercially available since then are not considered investigational studies)
16. Septicemia at the time of randomization/enrollment
17. Presence of other hemodynamically significant outflow lesions in the target limb requiring intervention at the time of the index procedure
18. Presence of aneurysm in the target vessel
19. Acute ischemia and/or acute thrombosis of the SFA/PPA prior to randomization/enrollment
20. Perforated vessel as evidenced by extravasation of contrast media prior to randomization/enrollment
21. Heavily calcified lesions
22. As applicable by French law, subject who is a protected individual such as an incompetent adult or incarcerated person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 775 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Torsello, MD, Principal Investigator — Sint-Franziskus-Hospital GmbH; Yann Goueffic, Principal Investigator — Hôpital St Joseph Paris
Locations (60):
- Austria (3):
  - LKH Innsbruck, Innsbruck
  - Klinikum Klagenfurt, Klagenfurt
  - Allgemeines Krankenhaus Wien, Vienna
- Belgium (8):
  - OLV Aalst, Aalst
  - ZiekenhuisNetwerk Antwerpen, Antwerp
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Regionaal Ziekenhuis Heilig Hart Tienen, Tienen
- France (13):
  - Hopital Privé Paul D'Egine, Champigny-sur-Marne
  - CHU - Hopital Gabriel Montpied, Clermont-Ferrand
  - L'Hôpital Henri-Mondor, Créteil
  - CHU Dijon, Dijon
  - CHU Lille, Lille
  - Hopital Edouard Herriot, Lyon
  - CHU Nancy, Nancy
  - Hopital Nord Laennec, Nantes
  - (Hôpital Européen Georges-Pompidou, Paris
  - CH de Saint-Nazaire, Saint-Nazaire
  - CHU Strasbourg, Strasbourg
  - Clinique Pasteur, Toulouse
  - CH Valenciennes, Valenciennes
- Germany (19):
  - Universitäts Herzzentrum, Bad Krozingen
  - Sankt Gertrauden-Krankenhaus, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Essen, Essen
  - Krankenhäuser Landkreis Freudenstadt GmbH, Freudenstadt
  - Universitätsklinikum Heidelberg, Heidelberg
  - SRH Klinikum Karlsbad-Langensteinbach, Karlsbad
  - University Hospital Schleswig-Holstein Campus Kiel, Kiel
  - University Medical Center of Johannes Gutenberg-Mainz, Mainz
  - Universitätsklinikum Marburg, Marburg
  - Klinik Diakoniewerk München-Maxvorstadt, München
  - St. Franziskus-Hospital Muenster, Münster
  - Universitätsklinikum Münster, Münster
  - Krankenhaus Barmherzige Brüder, Regensburg
  - RoMed Klinikum Rosenheim, Rosenheim
  - MEDINOS Kliniken Sonneberg GmbH, Sonneberg
  - Krankenhaus Torgau, Torgau
  - University Hospital of Tübingen, Tübingen
  - Klinikum Nordoberpfalz AG, Klinikum Weiden, Weiden
- Beaumont Hospital, Dublin, Ireland
- Italy (3):
  - San Raffaele Hospital, Milan
  - Centro cardiologico Monzino, Milan
  - Ospedaliero Universitaria Federico II, Naples
- Netherlands (2):
  - Hagaziekenhuis, The Hague
  - Elisabeth Tilburg Ziekenhuis, Tilburg
- Hospital Virgen Macarena, Seville, Spain
- Switzerland (2):
  - Inselspital Bern, Bern
  - Kantonsspital Luzern, Lucerne
- United Kingdom (8):
  - Royal Bournemouth Hospital, Bournemouth
  - Addenbrookes Hospital, Cambridge
  - Royal London Hospital, London
  - St.Thomas' Hospital, London
  - St. Mary's Hospital, London
  - Manchester University NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goueffic Y, Torsello G, Zeller T, Esposito G, Vermassen F, Hausegger KA, Tepe G, Thieme M, Gschwandtner M, Kahlberg A, Schindewolf M, Sapoval M, Diaz-Cartelle J, Stavroulakis K; EMINENT Investigators. Efficacy of a Drug-Eluting Stent Versus Bare Metal Stents for Symptomatic Femoropopliteal Peripheral Artery Disease: Primary Results of the EMINENT Randomized Trial. Circulation. 2022 Nov 22;146(21):1564-1576. doi: 10.1161/CIRCULATIONAHA.122.059606. Epub 2022 Oct 18. PMID 36254728

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Over an enrollment period of 41 months, 775 subjects were enrolled in the study of which, 508 subjects were enrolled in the investigational test device arm and 267 were enrolled in the bare metal stent (control device).
Groups:
- ELUVIA Stent Implantation: Percutaneous stent placement in the SFA/PPA
  ELUVIA (Stent Implantation): Drug-eluting self-expanding stent implantation during the index procedure.
- Control Bare Metal Stent Implantation: Percutaneous stent placement in the SFA/PPA of commercially available stents in Europe
  Permitted stents are Supera (Abbott), Lifestent (CR Bard), Everflex (Covidien/Medtronic), S.M.A.R.T. Flex (Cordis/Cardinal), S.M.A.R.T. Control (Cordis/Cardinal), Pulsar (Biotronik), COMPLETE SE (Medtronic), Misago (Terumo) or Innova (Boston Scientific)
Period: Overall Study
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Started | 508 | 267
Completed | 453 | 249
Not Completed | 55 | 18
Not completed — Withdrawal by Subject | 20 | 8
Not completed — Death | 12 | 3
Not completed — Protocol Violation | 17 | 6
Not completed — Early completion | 5 | 1
Not completed — Pending data entry | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation | Total
Number analyzed (Participants) | 508 | 267 | 775
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (8.7) | 68.9 (9.1) | 68.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 87 | 232
  Male | 363 | 180 | 543
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Black of African Heritage | 1 | 2 | 3
  Caucasian | 434 | 234 | 668
  Hispanic or Latino | 1 | 1 | 2
  Other | 16 | 8 | 24
  Not Disclosed | 55 | 21 | 76
Region of Enrollment [Number; unit: participants]
  Austria | 53 | 28 | 81
  Netherlands | 13 | 6 | 19
  Belgium | 71 | 40 | 111
  Ireland | 1 | 1 | 2
  Italy | 45 | 24 | 69
  United Kingdom | 15 | 10 | 25
  France | 73 | 34 | 107
  Switzerland | 18 | 12 | 30
  Germany | 206 | 106 | 312
  Spain | 13 | 6 | 19
History of Smoking [Count of Participants; unit: Participants]
  Current | 183 | 96 | 279
  Never | 91 | 44 | 135
  Previous | 201 | 111 | 312
  Unknown | 33 | 16 | 49
Current Diabetes Mellitus [Count of Participants; unit: Participants] | 180 | 96 | 276
History of Hyperlipidemia requiring medication [Count of Participants; unit: Participants] | 341 | 182 | 523
History of Hypertension requiring medication [Count of Participants; unit: Participants] | 397 | 203 | 600
History of Chronic Obstructive Pulmonary Disease [Count of Participants; unit: Participants] | 65 | 33 | 98
History of Coronary Artery Disease [Count of Participants; unit: Participants] | 159 | 96 | 255
History of Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 75 | 41 | 116
History of Congestive Heart Failure [Count of Participants; unit: Participants] | 35 | 13 | 48
History of Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 114 | 67 | 181
History of Coronary Artery Bypass Graft (CABG) Surgery [Count of Participants; unit: Participants] | 50 | 30 | 80
Current Anginal Status [Count of Participants; unit: Participants]
  Stable Angina | 19 | 7 | 26
  None | 482 | 250 | 732
  Unknown | 7 | 10 | 17
  Unstable Angina | 0 | 0 | 0
History of Transient Ischemic Attacks (TIA) [Count of Participants; unit: Participants] | 29 | 11 | 40
History of Cerebrovascular Accident (CVA) [Count of Participants; unit: Participants] | 38 | 15 | 53
History of Renal Insufficiency [Count of Participants; unit: Participants] | 59 | 22 | 81
History of Renal Percutaneous Intervention [Count of Participants; unit: Participants] | 6 | 5 | 11
History of Endovascular Interventions in Target Vessel [Count of Participants; unit: Participants] | 36 | 25 | 61
History of Other Peripheral Endovascular Interventions (other than Target Vessel) [Count of Participants; unit: Participants] | 147 | 86 | 233
History of Claudication [Count of Participants; unit: Participants] | 447 | 228 | 675

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Primary Patency at 12 Months Post-procedure
Description: The primary effectiveness endpoint assesses primary patency at 12 months post-procedure. This effectiveness endpoint is designed to demonstrate that the 12-month primary patency for the ELUVIA treatment group is superior to the Self-Expanding Bare Nitinol Stents treatment group.
Time Frame: 12 Months
Population: Primary patency defined as core-lab assessed duplex ultrasound peak systolic velocity ratio (PSVR) ≤ 2.4 at 12 months in the absence of clinically-driven Target Lesion Revascularization (TLR) or bypass of the target lesion.
  405/508 subjects in Eluvia and 222/267 subjects in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 405 | 222
Participants | 337 | 165
Statistical Analysis 1: Comparison: ELUVIA Stent Implantation vs Control Bare Metal Stent Implantation; Test type: Superiority; p = 0.0077, Chi-squared

2. Secondary Outcome: Number of Subjects Walking Improvement - Distance at Baseline to 12 Months
Description: Walking Improvement will be assessed and compared between the 2 study arms, by evaluating the change in Six Minute Hall Walk (6MHW) / treadmill test from baseline, or preceding any Target Vessel Revascularization and evaluating change in Walking Impairment Questionnaire (WIQ) from baseline.
  Values are represented as a mean and standard deviation and reflect the change in meters walked.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 508 | 267
Meter
  Baseline | 258.4 (153.4) | 239.1 (150.0)
  12 Month | 392.4 (286.0) | 361.9 (176.2)

3. Secondary Outcome: Number of Subjects Change in Quality of Life - Improvement From Baseline to 12 Month
Description: The change in quality of life will be assessed and compared between the 2 study arms, by evaluating change in EuroQol (EQ) - 5 Dimensions (5D) - 5 Levels (5L) questionnaire (EQ-5D-5L™) from baseline, or preceding any Target Vessel Revascularization Values are presented as a count of subjects at 12-months and by the number of subjects analyzed.
Time Frame: 12 Months
Population: The number analyzed for each row is based on the number of subjects that completed the portion of the quality-of-life assessment during the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 445 | 246
Participants
  Mobility Improvement: number analyzed (Participants) | 444 | 246
  Mobility Improvement | 295 | 158
  Self-Care Improvement | 39 | 19
  Usual Activities Improvement | 169 | 91
  Pain/ Discomfort Improvement: number analyzed (Participants) | 444 | 246
  Pain/ Discomfort Improvement | 238 | 143
  Anxiety/ Depression Improvement: number analyzed (Participants) | 444 | 246
  Anxiety/ Depression Improvement | 100 | 49

4. Secondary Outcome: Cost Effectiveness
Description: Cost effectiveness of ELUVIA™ drug-eluting stent versus bare metal self-expanding nitinol stents.
Time Frame: during index procedure, 1, 6, 12, 24 and 36 months
Population: Cost effectiveness was not collected for the study as this data was an optional health economics data analysis.
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Subjects With Clinical Improvement at 12-months
Description: Clinical improvement will be evaluated by assessing the changes in Rutherford Classification from baseline.
  Values are presented as a count of participants at 12-months by the number of participants analyzed.
  Rutherford Classification describes 7 categories of peripheral artery disease, including both the patient's clinical symptoms as well as objective findings;
  Primary sustained clinical improvement, is a rate of improvement in Rutherford classification of one or more categories as compared to baseline without the need for repeat target lesion revascularization (TLR);
  Secondary sustained clinical improvement is a rate of improvement in Rutherford classification of one or more categories as compared to baseline including those subjects with repeat TLR;
  Clinical deterioration, is the rate of downgrade in Rutherford classification of one or more categories as compared to baseline
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 440 | 244
Participants
  Primary Sustained Clinical Improvement - Improvement in Rutherford Classification without TLR | 365 | 187
  Secondary Sustained Clinical Improvement - Improvement in Rutherford Classification with TLR | 396 | 211
  No Change from Baseline | 40 | 30
  Clinical Deterioration | 4 | 3

6. Secondary Outcome: Number of Subjects With Hemodynamic Improvement at 12-months
Description: Hemodynamic improvement was evaluated by assessing the number of participants that demonstrated an increase in the Ankle-Brachial Index value of >/= 0.10 or an increase in the overall ABI value to >/= 0.90 from baseline to 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 419 | 233
Participants
  Hemodynamic Improvement | 331 | 179
  Hemodynamic Improvement - Including TLR | 355 | 196

7. Other Pre Specified Outcome: Number of Subjects With Walking Improvement at 1-month, 6-months, 12-months, 24-months, and 36-months
Description: Walking Improvement at 1-month, 6-months, 12-months, 24-months, and 36-months assessed by change in Walking Impairment Questionnaire (WIQ) from baseline.
Time Frame: 1, 6, 12, 24, and 36 months
Population: The number analyzed for each row is based on the number of subjects that completed the assessment during the specified visit.
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 508 | 267
Participants
  1 Month - PAD Specific Question - Number of Subjects Improved: number analyzed (Participants) | 346 | 190
  1 Month - PAD Specific Question - Number of Subjects Improved | 297 | 158
  1 Month - Distance Score - Number of Subjects Improved: number analyzed (Participants) | 334 | 185
  1 Month - Distance Score - Number of Subjects Improved | 299 | 162
  1 Month - Speed Scores - Number of Subjects Improved: number analyzed (Participants) | 317 | 177
  1 Month - Speed Scores - Number of Subjects Improved | 270 | 140
  1 Month - Stair Climbing Scores - Number of Subjects Improved: number analyzed (Participants) | 326 | 178
  1 Month - Stair Climbing Scores - Number of Subjects Improved | 238 | 133
  6 Month - PAD Specific Question - Number of Subjects Improved: number analyzed (Participants) | 446 | 243
  6 Month - PAD Specific Question - Number of Subjects Improved | 366 | 195
  6 Month - Distance Score - Number of Subjects Improved: number analyzed (Participants) | 438 | 239
  6 Month - Distance Score - Number of Subjects Improved | 381 | 216
  6 Month - Speed Scores - Number of Subjects Improved: number analyzed (Participants) | 419 | 229
  6 Month - Speed Scores - Number of Subjects Improved | 335 | 180
  6 Month - Stair Climbing Scores - Number of Subjects Improved: number analyzed (Participants) | 428 | 231
  6 Month - Stair Climbing Scores - Number of Subjects Improved | 309 | 164
  12 Month - PAD Specific Question - Number of Subjects Improved: number analyzed (Participants) | 438 | 241
  12 Month - PAD Specific Question - Number of Subjects Improved | 360 | 184
  12 Month - Distance Score - Number of Subjects Improved: number analyzed (Participants) | 434 | 237
  12 Month - Distance Score - Number of Subjects Improved | 372 | 204
  12 Month - Speed Scores - Number of Subjects Improved: number analyzed (Participants) | 412 | 225
  12 Month - Speed Scores - Number of Subjects Improved | 321 | 173
  12 Month - Stair Climbing Scores - Number of Subjects Improved: number analyzed (Participants) | 426 | 227
  12 Month - Stair Climbing Scores - Number of Subjects Improved | 300 | 159
  24 Month - PAD Specific Question - Number of Subjects Improved: number analyzed (Participants) | 402 | 223
  24 Month - PAD Specific Question - Number of Subjects Improved | 317 | 170
  24 Month - Distance Score - Number of Subjects Improved: number analyzed (Participants) | 396 | 219
  24 Month - Distance Score - Number of Subjects Improved | 344 | 188
  24 Month - Speed Scores - Number of Subjects Improved: number analyzed (Participants) | 376 | 204
  24 Month - Speed Scores - Number of Subjects Improved | 289 | 149
  24 Month - Stair Climbing Scores - Number of Subjects Improved: number analyzed (Participants) | 387 | 213
  24 Month - Stair Climbing Scores - Number of Subjects Improved | 269 | 143
  36 Month - PAD Specific Question - Number of Subjects Improved: number analyzed (Participants) | 375 | 216
  36 Month - PAD Specific Question - Number of Subjects Improved | 298 | 164
  36 Month - Distance Score - Number of Subjects Improved: number analyzed (Participants) | 373 | 215
  36 Month - Distance Score - Number of Subjects Improved | 304 | 178
  36 Month - Speed Scores - Number of Subjects Improved: number analyzed (Participants) | 352 | 201
  36 Month - Speed Scores - Number of Subjects Improved | 256 | 135
  36 Month - Stair Climbing Scores - Number of Subjects Improved: number analyzed (Participants) | 365 | 206
  36 Month - Stair Climbing Scores - Number of Subjects Improved | 243 | 123

8. Other Pre Specified Outcome: Number of Subjects With Quality of Life Improvement at 1-month, 6-months, 24-months, and 36-months
Description: Quality of Life Improvement will be assessed at 1-month, 6-months, 24-months, and 36-months by evaluating the change in EQ-5D-5L™ from baseline
Time Frame: 1, 6, 24, and 36 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 508 | 267
Participants
  1 Month - Mobility Improvement: number analyzed (Participants) | 351 | 192
  1 Month - Mobility Improvement | 257 | 137
  1 Month - Self Care Improvement: number analyzed (Participants) | 351 | 192
  1 Month - Self Care Improvement | 30 | 11
  1 Month - Usual Activities Improvement: number analyzed (Participants) | 351 | 192
  1 Month - Usual Activities Improvement | 130 | 76
  1 Month - Pain/ Discomfort Improvement: number analyzed (Participants) | 350 | 192
  1 Month - Pain/ Discomfort Improvement | 217 | 120
  1 Month - Anxiety/ Depression Improvement: number analyzed (Participants) | 350 | 190
  1 Month - Anxiety/ Depression Improvement | 70 | 35
  6 Month - Mobility Improvement: number analyzed (Participants) | 452 | 247
  6 Month - Mobility Improvement | 307 | 162
  6 Month - Self Care Improvement: number analyzed (Participants) | 452 | 247
  6 Month - Self Care Improvement | 41 | 18
  6 Month - Usual Activities Improvement: number analyzed (Participants) | 452 | 247
  6 Month - Usual Activities Improvement | 168 | 95
  6 Month - Pain/ Discomfort Improvement: number analyzed (Participants) | 452 | 247
  6 Month - Pain/ Discomfort Improvement | 258 | 142
  6 Month - Anxiety/ Depression Improvement: number analyzed (Participants) | 450 | 245
  6 Month - Anxiety/ Depression Improvement | 86 | 53
  24 Month - Mobility Improvement: number analyzed (Participants) | 408 | 228
  24 Month - Mobility Improvement | 269 | 148
  24 Month - Self Care Improvement: number analyzed (Participants) | 408 | 228
  24 Month - Self Care Improvement | 32 | 18
  24 Month - Usual Activities Improvement: number analyzed (Participants) | 408 | 228
  24 Month - Usual Activities Improvement | 149 | 86
  24 Month - Pain/ Discomfort Improvement: number analyzed (Participants) | 408 | 228
  24 Month - Pain/ Discomfort Improvement | 211 | 137
  24 Month - Anxiety/ Depression Improvement: number analyzed (Participants) | 408 | 227
  24 Month - Anxiety/ Depression Improvement | 89 | 51
  36 Month - Mobility Improvement: number analyzed (Participants) | 378 | 221
  36 Month - Mobility Improvement | 238 | 136
  36 Month - Self Care Improvement: number analyzed (Participants) | 378 | 222
  36 Month - Self Care Improvement | 30 | 15
  36 Month - Usual Activities Improvement: number analyzed (Participants) | 378 | 221
  36 Month - Usual Activities Improvement | 136 | 78
  36 Month - Pain/ Discomfort Improvement: number analyzed (Participants) | 379 | 222
  36 Month - Pain/ Discomfort Improvement | 191 | 104
  36 Month - Anxiety/ Depression Improvement: number analyzed (Participants) | 378 | 222
  36 Month - Anxiety/ Depression Improvement | 76 | 42

9. Other Pre Specified Outcome: Number of Subjects With Clinical Improvement at 1-month, 6-months, 24-months, and 36-months
Description: Clinical improvement will be evaluated by assessing the changes in Rutherford Classification from baseline
Time Frame: 1, 6, 24, and 36 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 508 | 267
Participants
  1 Month - Primary Sustained Clinical Improvement: number analyzed (Participants) | 354 | 190
  1 Month - Primary Sustained Clinical Improvement | 328 | 175
  1 Month - Secondary Sustained Clinical Improvement: number analyzed (Participants) | 354 | 190
  1 Month - Secondary Sustained Clinical Improvement | 329 | 176
  1 Month - No Change from Baseline: number analyzed (Participants) | 354 | 190
  1 Month - No Change from Baseline | 22 | 13
  1 Month - Clinical Deterioration: number analyzed (Participants) | 354 | 190
  1 Month - Clinical Deterioration | 3 | 1
  6 Month - Primary Sustained Clinical Improvement: number analyzed (Participants) | 455 | 248
  6 Month - Primary Sustained Clinical Improvement | 403 | 223
  6 Month - Secondary Sustained Clinical Improvement: number analyzed (Participants) | 455 | 248
  6 Month - Secondary Sustained Clinical Improvement | 415 | 227
  6 Month - No Change from Baseline: number analyzed (Participants) | 455 | 248
  6 Month - No Change from Baseline | 35 | 17
  6 Month - Clinical Deterioration: number analyzed (Participants) | 455 | 248
  6 Month - Clinical Deterioration | 5 | 4
  24 Month - Primary Sustained Clinical Improvement: number analyzed (Participants) | 399 | 226
  24 Month - Primary Sustained Clinical Improvement | 304 | 170
  24 Month - Secondary Sustained Clinical Improvement: number analyzed (Participants) | 399 | 226
  24 Month - Secondary Sustained Clinical Improvement | 356 | 201
  24 Month - No Change from Baseline: number analyzed (Participants) | 399 | 226
  24 Month - No Change from Baseline | 35 | 24
  24 Month - Clinical Deterioration: number analyzed (Participants) | 399 | 226
  24 Month - Clinical Deterioration | 8 | 1
  36 Month - Primary Sustained Clinical Improvement: number analyzed (Participants) | 379 | 216
  36 Month - Primary Sustained Clinical Improvement | 263 | 152
  36 Month - Secondary Sustained Clinical Improvement: number analyzed (Participants) | 379 | 216
  36 Month - Secondary Sustained Clinical Improvement | 336 | 188
  36 Month - No Change from Baseline: number analyzed (Participants) | 379 | 216
  36 Month - No Change from Baseline | 35 | 22
  36 Month - Clinical Deterioration: number analyzed (Participants) | 379 | 216
  36 Month - Clinical Deterioration | 8 | 6

10. Other Pre Specified Outcome: Number of Subjects With Hemodynamic Improvement at 1-month, 6-months, 24-months, and 36-months
Description: The hemodynamic improvement will be evaluated by assessing changes in Ankle-Brachial Index (ABI) from baseline
Time Frame: 1, 6, 24, and 36 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 508 | 267
Participants
  1 Month - Hemodynamic Improvement: number analyzed (Participants) | 329 | 181
  1 Month - Hemodynamic Improvement | 287 | 163
  1 Month - Hemodynamic Improvement (Including TLR): number analyzed (Participants) | 329 | 181
  1 Month - Hemodynamic Improvement (Including TLR) | 288 | 164
  6 Month - Hemodynamic Improvement: number analyzed (Participants) | 432 | 239
  6 Month - Hemodynamic Improvement | 355 | 196
  6 Month - Hemodynamic Improvement (Including TLR): number analyzed (Participants) | 432 | 239
  6 Month - Hemodynamic Improvement (Including TLR) | 366 | 200
  24 Month - Hemodynamic Improvement: number analyzed (Participants) | 366 | 205
  24 Month - Hemodynamic Improvement | 248 | 145
  24 Month - Hemodynamic Improvement (Including TLR): number analyzed (Participants) | 366 | 205
  24 Month - Hemodynamic Improvement (Including TLR) | 293 | 166
  36 Month - Hemodynamic Improvement: number analyzed (Participants) | 346 | 190
  36 Month - Hemodynamic Improvement | 215 | 123
  36 Month - Hemodynamic Improvement (Including TLR): number analyzed (Participants) | 346 | 190
  36 Month - Hemodynamic Improvement (Including TLR) | 272 | 154

11. Other Pre Specified Outcome: Primary Patency and Assisted Primary Patency
Description: Primary Patency and Assisted Primary Patency at 6 months, 12 months using different Duplex Ultrasound (DUS) and Peak Systolic Velocity Ration (PSVRs). All DUS readings will be assessed by an independent core laboratory. Primary Patency is reported at 6 and 12-months.
Time Frame: 6 and 12 months
Population: The number analyzed indicates the subjects with available diagnostic duplex ultrasound images.
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 508 | 267
Participants
  6 Month - Primary Patency: number analyzed (Participants) | 434 | 228
  6 Month - Primary Patency | 395 | 195
  6 Month - Assisted Primary Patency: number analyzed (Participants) | 425 | 226
  6 Month - Assisted Primary Patency | 409 | 200
  12 Month - Primary Patency: number analyzed (Participants) | 405 | 222
  12 Month - Primary Patency | 337 | 165
  12 Month - Assisted Primary Patency: number analyzed (Participants) | 389 | 214
  12 Month - Assisted Primary Patency | 360 | 182

12. Other Pre Specified Outcome: Adverse Event and Major Adverse Event (MAE) Rate
Description: Adverse Event rate and Major Adverse Event rate, defined as all causes of death, target limb major amputation and/or Target Lesion Revascularization, rate at each time point
Time Frame: 1, 6, 12, 24, and 36 months
Population: The number Started in Participant Flow indicates the intent-to-treat population while the number analyzed indicates the as-treated (AT) population. For AT analysis, subjects implanted are included based on the actual Test or Control device each subject received (including cross-over subjects). Only study permitted stents are included in the AT set.
  The number analyzed in the data table differs from the overall analyzed as it indicates subjects that reached the lower limit for the visit window.
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 492 | 273
Participants
  1 Month Adverse Event Rate | 77 | 32
  6 Month Adverse Event Rate | 105 | 54
  12 Month Adverse Event Rate | 134 | 79
  24 Month Adverse Event Rate | 181 | 96
  36 Month Adverse Event Rate | 215 | 111
  1 Month - MAE - All Cause Death: number analyzed (Participants) | 489 | 272
  1 Month - MAE - All Cause Death | 3 | 0
  1 Month - MAE - Target Limb Major Amputation: number analyzed (Participants) | 489 | 272
  1 Month - MAE - Target Limb Major Amputation | 1 | 0
  1 Month - MAE - Target Lesion Revascularization: number analyzed (Participants) | 489 | 272
  1 Month - MAE - Target Lesion Revascularization | 2 | 2
  6 Month - MAE - All Cause Death: number analyzed (Participants) | 485 | 266
  6 Month - MAE - All Cause Death | 7 | 3
  6 Month - MAE - Target Limb Major Amputation: number analyzed (Participants) | 485 | 266
  6 Month - MAE - Target Limb Major Amputation | 1 | 0
  6 Month - MAE - Target Lesion Revascularization: number analyzed (Participants) | 485 | 266
  6 Month - MAE - Target Lesion Revascularization | 23 | 7
  12 Month - MAE - All Cause Death: number analyzed (Participants) | 474 | 263
  12 Month - MAE - All Cause Death | 13 | 3
  12 Month - MAE - Target Limb Major Amputation: number analyzed (Participants) | 474 | 263
  12 Month - MAE - Target Limb Major Amputation | 1 | 0
  12 Month - MAE - Target Lesion Revascularization: number analyzed (Participants) | 474 | 263
  12 Month - MAE - Target Lesion Revascularization | 42 | 28
  24 Month - MAE - All Cause Death: number analyzed (Participants) | 461 | 259
  24 Month - MAE - All Cause Death | 28 | 8
  24 Month - MAE - Target Limb Major Amputation: number analyzed (Participants) | 461 | 259
  24 Month - MAE - Target Limb Major Amputation | 1 | 0
  24 Month - MAE - Target Lesion Revascularization: number analyzed (Participants) | 461 | 259
  24 Month - MAE - Target Lesion Revascularization | 71 | 45
  36 Month - MAE - All Cause Death: number analyzed (Participants) | 451 | 255
  36 Month - MAE - All Cause Death | 38 | 15
  36 Month - MAE - Target Limb Major Amputation: number analyzed (Participants) | 451 | 255
  36 Month - MAE - Target Limb Major Amputation | 2 | 1
  36 Month - MAE - Target Lesion Revascularization: number analyzed (Participants) | 451 | 255
  36 Month - MAE - Target Lesion Revascularization | 100 | 53

13. Other Pre Specified Outcome: Clinically-driven Target Lesion Revascularization (TLR) Rate
Description: Target Lesion Revascularization, defined as any surgical or percutaneous intervention to the target lesion(s) after the index procedure, rate at each time point.
Time Frame: 1, 6, 12, 24, and 36 months
Population: The number started in participant flow indicates the intent-to-treat population while the number analyzed indicates the the as-treated population.
  For as-treated analysis, all subjects in the per-protocol population will be included based on the actual Test or Control device that each subject received (i.e. including cross-over subjects).
  The number analyzed in the rows below differs from the overall analyzed as it indicates the subjects that reached the lower limit for the visit window.
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 492 | 273
Participants
  1 Month - Clinically-driven TLR: number analyzed (Participants) | 489 | 272
  1 Month - Clinically-driven TLR | 3 | 2
  6 Month - Clinically-driven TLR: number analyzed (Participants) | 479 | 266
  6 Month - Clinically-driven TLR | 23 | 7
  12 Month - Clinically-driven TLR: number analyzed (Participants) | 474 | 263
  12 Month - Clinically-driven TLR | 40 | 28
  24 Month - Clinically-driven TLR: number analyzed (Participants) | 435 | 251
  24 Month - Clinically-driven TLR | 69 | 45
  36 Month - Clinically-driven TLR: number analyzed (Participants) | 417 | 244
  36 Month - Clinically-driven TLR | 97 | 53

14. Other Pre Specified Outcome: Clinically-driven Target Vessel Revascularization (TVR) Rate
Description: Target Vessel Revascularization, defined as any surgical or percutaneous intervention to the target vessel after the index procedure, rate at each time point.
Time Frame: 1, 6, 12, 24 and 36 months
Population: The number analyzed indicates the subjects that reached the lower limit for the visit window.
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 492 | 273
Participants
  1 Month - Clinically-driven TVR: number analyzed (Participants) | 489 | 272
  1 Month - Clinically-driven TVR | 4 | 4
  6 Month - Clinically-driven TVR: number analyzed (Participants) | 485 | 266
  6 Month - Clinically-driven TVR | 26 | 10
  12 Month - Clinically-driven TVR: number analyzed (Participants) | 474 | 263
  12 Month - Clinically-driven TVR | 52 | 30
  24 Month - Clinically-driven TVR: number analyzed (Participants) | 435 | 251
  24 Month - Clinically-driven TVR | 77 | 48
  36 Month - Clinically-driven TVR: number analyzed (Participants) | 417 | 244
  36 Month - Clinically-driven TVR | 105 | 56

15. Other Pre Specified Outcome: Technical Success
Description: Technical success defined as delivery and deployment of the assigned study stent to the target lesion to achieve residual angiographic stenosis no greater than 30% assessed visually
Time Frame: during index procedure after stent delivered and deployed to the target lesion
Population: The number started in participant flow indicates the intent-to-treat population while the number analyzed indicates the the as-treated population.
  For as-treated analysis, all subjects in the per-protocol population will be included based on the actual Test or Control device that each subject received (i.e. including cross-over subjects).
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 491 | 273
Participants | 488 | 269

16. Other Pre Specified Outcome: Procedural Success
Description: Procedural success defined as technical success with no MAEs noted within 24 hours of the index procedure
Time Frame: within 24 hours of stenting procedure
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 491 | 273
Participants | 488 | 269

17. Other Pre Specified Outcome: Number of Stent Fractures
Description: Number of Stent Fractures reported at 12 months utilizing the Vascular InterVentional Advances (VIVA) definitions assessed by an independent core laboratory.
  Stent fractures were analyzed if sites collected imaging per standard of care (SOC).
Time Frame: 12 Months
Measure: Count of Units; unit: Stents
Units Other Than Participants: Stents
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
Number analyzed (Participants) | 508 | 267
Number analyzed (Stents) | 21 | 16
Stents | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 36 months follow up.
Description: All-cause mortality is analyzed for the ITT population. Safety endpoints included SAE and Other (not Including Serious) Adverse Events, is analyzed for the As-treated (AT) population.
  Subjects who receive either ELUVIA or bare metal stents (BMS) at procedure are included in the AT analysis set according to the treatment actually received (even if not the treatment they were randomized to). Subjects who do not receive ELUVIA or study permitted BMS are excluded from the AT analysis set.
Arm/Group | ELUVIA Stent Implantation | Control Bare Metal Stent Implantation
All-Cause Mortality (participants affected / at risk) | 39/508 | 15/267
Serious Adverse Events (participants affected / at risk) | 181/492 | 90/273
Other Adverse Events (participants affected / at risk) | 109/492 | 54/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELUVIA Stent Implantation (N=492) | Control Bare Metal Stent Implantation (N=273)
Peripheral artery occlusion (Vascular disorders) | 32 (40) | 5 (6)
Peripheral artery stenosis (Vascular disorders) | 32 (38) | 17 (19)
Intermittent claudication (Vascular disorders) | 11 (12) | 3 (3)
Peripheral ischaemia (Vascular disorders) | 5 (5) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (4) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 1 (1)
Peripheral embolism (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Reperfusion injury (Vascular disorders) | 1 (1) | 0 (0)
Vascular dissection (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery dissection (Vascular disorders) | 0 (0) | 2 (2)
Vascular stent restenosis (General disorders) | 21 (21) | 19 (28)
Vascular stent thrombosis (General disorders) | 12 (14) | 6 (6)
Vascular stent stenosis (General disorders) | 10 (11) | 10 (11)
Death (General disorders) | 11 (11) | 6 (6)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 1 (1) | 0 (0)
Stenosis (General disorders) | 1 (1) | 4 (4)
Device embolisation (General disorders) | 0 (0) | 1 (1)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 7 (7) | 4 (4)
Reocclusion (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 9 (9) | 9 (13)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 20 (23) | 6 (6)
Pneumonia (Infections and infestations) | 6 (6) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Venous stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vascular stent occlusion (General disorders) | 9 (11) | 2 (2)
Catheter site inflammation (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELUVIA Stent Implantation (N=492) | Control Bare Metal Stent Implantation (N=273)
Peripheral artery stenosis (Vascular disorders) | 11 (13) | 7 (7)
Peripheral artery occlusion (Vascular disorders) | 11 (12) | 5 (5)
Haematoma (Vascular disorders) | 5 (5) | 4 (4)
Vascular dissection (Vascular disorders) | 4 (4) | 0 (0)
Femoral artery dissection (Vascular disorders) | 3 (3) | 6 (6)
Artery dissection (Vascular disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Arterial spasm (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular occlusion (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenus fistula (Vascular disorders) | 0 (0) | 1 (1)
Vascular stent restenosis (General disorders) | 9 (9) | 12 (12)
Vascular stent stenosis (General disorders) | 5 (5) | 4 (4)
Vessel puncture site haematoma (General disorders) | 4 (4) | 3 (3)
Vascular stent thrombosis (General disorders) | 5 (5) | 1 (1)
Stenosis (General disorders) | 2 (2) | 2 (2)
Puncture site haemorrhage (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Puncture site pain (General disorders) | 1 (1) | 0 (0)
Device embolisation (General disorders) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 10 (10) | 2 (2)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 6 (6) | 5 (5)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin maceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Contrast media reaction (Immune system disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 7 (7) | 0 (0)
Vascular stent occlusion (General disorders) | 7 (7) | 0 (0)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
COVID-19 pandemic impacted the amount of imaging data collected causing insufficiencies to calculate rates to appropriately report some outcome measures particularly with data at 24 and 36 months follow up visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Protocol (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT02921230/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT02921230/SAP_001.pdf